CLINICAL TRIAL: NCT00780637
Title: Characterization of Brachial Arterial t-PA Release, Vasodilator Function, and Vascular Compliance and Correlation With Fibrinolytic Balance, Oxidative Stress, and Inflammation Measures in Heart Transplant Recipients (SCCOR Project 1, Aim 3C)
Brief Title: Brachial Artery t-PA Release in Heart Transplant Recipients
Acronym: P1A3C
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Bradykinin Shortage, SCCOR expired prior to BK availability, lack of enrollment.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, James Muldowney, Assistant Professor of Medicine, Vanderbilt University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 070517
Expanded Access: Available
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Heart Transplantation
Keywords: Heart Transplant; Endothelial Function; Fibrinolysis; Transplant recipients at baseline
MeSH Terms: interventions — Bradykinin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bradykinin (Experimental): Patients receive 0, 10, 20, and 40 ng/min/100cc forearm volume of intrabrachial bradykinin, for 5 minutes at each dose. Forearm blood flow will be measured by strain gauge plethysmography, blood samples will be obtained to measure t-PA, PAI-1 at each dose. FMD and Radial artery tonometry will also be performed under resting conditions.
  Interventions: Drug: Bradykinin

INTERVENTIONS:
Drug: Bradykinin — Patients receive 0, 10, 20, and 40 ng/100cc forearm volume/min of bradykinin intrabrachial.

SUMMARY:
Bradykinin stimulates t-PA release from intact vessels, but not from endothelial cells in culture. It has been proposed that the nerves of blood vessels are the source of bradykinin stimulated t-PA release. In order tho test this hypothesis, we intend to infuse bradykinin into the brachial (arm) artery and the coronary arteries of heart transplant recipients and control subjects. This is because heart transplant recipients do not have nerves to their coronary arteries.

This protocol studies the effects of bradykinin on t-PA release in the forearm of transplant recipients. The brachial artery has intact nerves.

Separate protocols address coronary artery infusions in healthy subjects and transplant recipients and forearm infusions in healthy subjects.

ELIGIBILITY:
Inclusion criteria:

1. Adults 18 years and greater who have undergone heart transplantation
2. Healthy

Exclusion criteria:

1. PVC < 30
2. Hypertensive subjects on ACE inhibitors
3. Pregnant or nursing mothers
4. Diabetic with HbA1C > 7.5 or stigmata of end organ damage (neuropathy, retinopathy, nephropathy, cardiomyopathy)
5. Cholesterol > 30 mg/dL above NCEP accepted level based on cardiac risk.
6. Triglycerides > 200
7. Previously diagnosed obstructive coronary artery disease
8. Renal insufficiency (Creatinine ≥ 1.5 mg/dl)
9. History of cerebrovascular disease
10. Any chronic inflammatory disease (rheumatologic, inflammatory bowel disease, etc)
11. Uncontrolled Stage 2 Hypertension (160/100 mmHg), or end organ damage due to hypertension (left ventricular hypertrophy, atrial fibrillation, hematuria, renal insufficiency, prior cerebrovascular disease).
12. Angiotensin converting enzyme inhibitor use
13. Coagulopathy (INR ≥ 1.5, PTT ≥ 150% of control)
14. Peripheral Vascular Disease
15. Other chronic medical illnesses at the discretion of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Peak t-PA release | Single Study Visit

SECONDARY OUTCOMES:
t-PA release at various doses | Single Study Visit

CONTACTS AND LOCATIONS:
Overall Officials: James AS Muldowney, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States